CLINICAL TRIAL: NCT00996944
Title: Clinical Evaluation of Ropinirole IR (Immediate Release) Tablets in Patients Who Are Diagnosed With Symptomatic Restless Legs Syndrome (RLS) Associated With Chronic Kidney Disease (CKD) Managed With Haemodialysis (Including Haemofiltration and Haemodiafiltration)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Because GSK concluded that it was impossible to recruit sufficient participants within a reasonable timeframe.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113079
Record Dates: First submitted 2009-10-08; First posted 2009-10-16 (Estimated); Results first posted 2011-06-13 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-06

CONDITIONS: Restless Legs Syndrome
Keywords: ropinirole; haemodialysis; restless legs syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ropinirole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropinirole IR (Experimental)
  Interventions: Drug: Ropinirole immediate release (IR)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropinirole immediate release (IR) — Subjects completing the screening period will be randomized (1:1) to receive the IR or placebo for 12 weeks. The treatment will be started at the initial dose of 0.25 mg/day within 1 to 3 hours before bedtime. The maximum available dose is 3 mg/day. For all subjects completing short-term period and entering the long-term treatment period, the open-label treatment will be started from IR 0.25 mg/ day regardless of dose levels during short-term period. The dose will be upward titrated from 0.25 mg/day to 0.5 mg/day and after that in increments of 0.5 mg/day until sufficient efficacy is obtained (targeting "much improved" or "very much improved" in the CGI-I) without safety/tolerability problem.
  Arms: Ropinirole IR
Drug: Placebo — Subjects completing the screening period will be randomized (1:1) to receive the IR or placebo for 12 weeks. The treatment will be started at the initial dose of 0.25 mg/day within 1 to 3 hours before bedtime.
  Arms: Placebo

SUMMARY:
This is a multicenter, placebo controlled, parallel group, double-blind, randomized comparison study to evaluate the efficacy and safety of ropinirole IR tablets orally administered for 12 weeks in patients with symptomatic restless legs syndrome associated with Chronic kidney disease (CKD) managed with haemodialysis (including haemofiltration and haemodiafiltration) (hereinafter referred to as "uRLS"), to evaluate the efficacy and safety of long-term administration of ropinirole IR tablets, and assess the effect on the steady state pharmacokinetics in the long-term administration period of ropinirole IR tablets.

ELIGIBILITY:
Inclusion Criteria:

at Week -1 (at the screening visit)

* Patients who are diagnosed with symptomatic restless legs syndrome associated with Chronic kidney disease (CKD) managed with haemodialysis (including haemofiltration and haemodiafiltration). RLS are diagnosed based on the International RLS Study Group's (IRLSSG) Diagnostic Criteria.
* Patients with chronic kidney disease (CKD) on haemodialysis (including haemofiltration and haemodiafiltration) for at least 3 months prior to the screening period with and receiving an adequate haemodialysis prescription (i.e. single-pool Kt/V >1.0. Shinzato calculating formula [Shinzato, 1994] using in Japanese Society for Dialysis Therapy will be used.)
* Patients aged ≥18 years and <80 years.
* Patients who have had RLS symptoms for 20 days or more on or after 28 days before the start of the screening period. However, patients who have been receiving drug therapy for RLS before the start of the screening period do not apply to this criterion when meeting the conditions below: The patient's drug therapy (excluding Anxiolytics and Hypnotics and sedatives medication) for RLS can be discontinued at the time of starting the screening period. For RLS symptoms in the subject was considered to have continued for 20 days or more on or after 28 days before the start of the drug treatment for RLS.
* QTc criteria (QTc [b or f], mechanical or manual reread, male or female): Patients with QTc <450 msec or <480 msec for patients with bundle branch block (BBB) -values based on either single electrocardiogram (ECG) values or triplicate ECG averaged QTc values obtained over a brief recording period.
* Male or female patients. A female subject is eligible to enter and participate in the study if she:

Is of non-childbearing potential or Is of child-bearing potential, is not lactating and agrees to use one of GlaxoSmithKline (GSK)-specified highly effective methods for avoiding pregnancy: abstinence, oral contraceptives, either combined or progestogen alone (see "Permitted medications"), injectable progestogen, implants of levonorgestrel, estrogenic vaginal ring (see "Permitted medications"), percutaneous contraceptive patches (see "Permitted medications"), intrauterine device (IUD) or intrauterine system (IUS) that meets the SOP effectiveness criteria as stated in the product label, male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject, double barrier method (condom or occlusive cap [diaphragm or cervical/vault caps] plus spermicidal agent [foam/gel/film/cream/suppository]).

* Outpatients
* Patients who are able to give informed written consent in person. Legal representative also should give informed written consent, if patients are under twenty years old.

at Week 0 (at the start of the treatment period)

* Patients who experience RLS symptoms for at least 4 days within 7 days before the start of the treatment period.
* Patients who have sleep disturbance associated with RLS. Patients who answered as 3 (severe) or 4 (very severe) to Question 4 (Sleep disturbance) in the IRLS Rating Scale.
* Patients whose IRLS Rating Scale total scores are 15 points or more.
* Liver function tests: Patients with aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 * ULN (upper limit of normal); and bilirubin ≤ 1.5 * ULN (isolated bilirubin > 1.5 ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) at week -1(at the screening visit). ULN of ALT(GTP) and AST(GOT) is 20 IU/L [Kurokawa, 2002].
* A female subject has a negative pregnancy test at week -1(at the screening visit).

Exclusion Criteria:

at Week -1 (at the screening visit)

* Patients with signs of primary RLS (Patients who have developed RLS symptoms since kidney function was normal)
* Patients with following sleep disorder not associated with RLS e.g. narcolepsy, sleep terror disorder, sleepwalking disorder, breathing related sleep disorder
* Patients with complication of movement disorder (e.g. Parkinson's disease, dyskinesia, dystonia, etc)
* Patients with severe hepatic/cardiac/pulmonary disorder or haematopoietic disorder other than those on haemodialysis (including haemofiltration and haemodiafiltration). The severity refers to Grade 3 according to "the Classification of the Severity of Adverse Experiences" (Pharmaceutical affairs bureau/Safety division(PAB/SD) Notification No. 80, dated 29 June 1992).
* Patients with a history of malignancies within the past 5 years, with the exception of basal cell carcinoma of the skin or carcinoma in situ of cervix.
* Patients with a medical history or complication of substance abuse (e.g. alcohol or drug) or dependency of substance for the last one year.
* Patients with supine systolic blood pressure (SBP) of <100 mmHg or >190 mmHg or supine diastolic blood pressure (DBP) of ≥120 mmHg before the dialysis which will be conducted after the longest interval,at the screening visit.
* Patients intolerant to ropinirole hydrochloride (HCl) or other dopamine agonists.
* Patients for whom ropinirole HCl or other dopamine agonists are considered to be of safety concern by the investigator/subinvestigator
* Patients with a history of augmentation or End-of-dose-rebound in the early morning after medications of dopamine agonists (including ropinirole HCl) and/or L-Dopa. Augmentation is defined as follows: RLS symptoms that occurred while on treatment and occur ≧ 2 hours earlier than they did before. Symptoms which are more severe than when not treated. Symptoms which start after less time at rest than they did before treatment. Symptoms which involve other parts of the body, such as the arms or trunk.
* Patients without night time sleeping habit (e.g. night-shift worker, etc) and those who must drastically change the habitual bedtime during the study duration.
* Patients who have participated in another clinical study of an investigational product or medical device within the last 12 weeks prior to the start of the screening period.
* Female patients who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study. (Instructions should be given to women of childbearing potential to practice adequate contraception even if they have no plan for pregnancy).
* Current or chronic history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Presence of hepatitis B surface antigen (HBsAg), positive Hepatitis C test result within 3 months of screening.
* Patients who have medical conditions which, in the opinion of investigator/subinvestigator could affect efficacy and safety assessment. This may include the following disorders: fibromyalgia syndrome, rheumatoid arthritis, symptomatic orthostatic hypotension, hepatic failure, pulmonary fibrosis.
* Subject is unable to discontinue prohibited medications during the Screening period.
* Subjects who know they will imminently receive a transplant
* Patients who have changed the dose or administration method of Anxiolytics or Hypnotics and sedatives within the last 4 weeks prior to the start of the screening period and or Patients who used more than two drugs.
* Others whom the investigator/subinvestigator considers ineligible for the study.

at Week 0 (start of the treatment period)

* Patients with supine SBP of <100 mmHg or >190 mmHg or supine DBP of ≥120 mmHg before the dialysis which will be conducted after the longest interval, at Week 0 (start of the treatment period).
* Patients who have started treatment with medications including an estrogen drug product, a drug that is known to substantially induce or inhibit CYP1A2, an antihistamine (for ocular instillation or dermal application, or a preparation containing fexofenadine HCl or loratadine), Anxiolytics, Hypnotics and sedatives or who have changed the dose or administration method of such medications between Week -1 (start of the screening period) and Week 0 (start of the treatment period).
* Patients whose serum ferritin level is <10 μg/L (ng/mL) at the screening visit.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-11-30; Primary Completion 2010-06-01 (Actual); Study Completion 2010-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Japan (15):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokushima

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113079 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113079 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113079 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113079 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was prematurely terminated after 5 months had passed since its initiation, because GlaxoSmithKline (GSK) concluded that it was impossible to recruit sufficient participants within a reasonable timeframe. In this study, no participants had completed. The maximum duration was 24 weeks plus follow-up (up to Week 64).
Groups:
- Ropinirole IR-Ropinirole IR: Participants received immediate-release (IR) tablets of ropinirole once daily for 12 weeks in the double-blind treatment period. The dose of investigational product (IP) was upward titrated from 0.25 milligrams (mg)/day to 0.5 mg/day at an interval of at least 1 week, followed by upward titration in increments of 0.5 mg/day at intervals of at least 1 week until sufficient efficacy was obtained (targeting "much improved" or "very much improved" in the investigator/subinvestigator-assessed Clinical Global Impression-Improvement [CGI-I]) without a safety/tolerability problem, although the dose did not exceed 3 mg/day. All participants completing the double-blind treatment period were eligible to continue in the open-label long-term treatment period. In the open-label period, participants were to receive ropinirole IR tablets once daily for 52 weeks with a similar upward titration method as in the double-blind treatment period.
- Placebo-Ropinirole IR: Participants received matching placebo to ropinirole IR in the double-blind treatment period. All participants completing the double-blind treatment period were eligible to continue in the open-label long-term treatment period. In the open-label period, participants received ropinirole IR tablets in the same way as in the ropinirole IR-ropinirole IR group.
Period: Double-blind Treatment Period
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Started | 22 | 12
Completed | 12 | 5
Not Completed | 10 | 7
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Study Closed/Terminated | 6 | 5
Not completed — Withdrawal by Subject | 1 | 1
Period: Long-term Treatment Period
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Started | 12 | 5
Completed | 0 | 0
Not Completed | 12 | 5
Not completed — Study Closed/Terminated | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Ropinirole IR-Ropinirole IR: Participants received immediate-release (IR) tablets of ropinirole once daily for 12 weeks in the double-blind treatment period. The dose of investigational product (IP) was upward titrated from 0.25 milligram (mg)/day to 0.5 mg/day at an interval of at least 1 week, followed by upward titration in increments of 0.5 mg/day at intervals of at least 1 week until sufficient efficacy was obtained (targeting "much improved" or "very much improved" in the investigator/subinvestigator-assessed Clinical Global Impression - Improvement [CGI-I]) without a safety/tolerability problem, although the dose did not exceed 3 mg/day. All participants completing the double-blind treatment period were eligible to continue in the open-label long-term treatment period. In the open-label period, participants were to receive ropinirole IR tablets once daily for 52 weeks with a similar upward titration method as in the double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR | Total
Number analyzed (Participants) | 22 | 12 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (11.39) | 53.8 (10.90) | 53.6 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 19 | 8 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - Japanese Heritage | 22 | 12 | 34
  Not Asian - Japanese Heritage | 0 | 0 | 0
Age at Onset of Restless Legs Syndrome [Mean (Standard Deviation); unit: years] | 48.9 (11.24) | 49.4 (10.12) | 49.1 (10.71)
Duration of Dialysis [Mean (Standard Deviation); unit: years] | 7.41 (5.537) | 6.08 (5.274) | 6.94 (5.403)

OUTCOME MEASURES:

1. Primary Outcome: International Restless Legs Syndrome (IRLS) Rating Scale Total Score at Week 0 and Week 12
Description: The IRLS rating scale is an investigator-rated scale consisting of 10 questions with a choice of 5 responses each. These responses are numerically scored from 0 (the least severe response) to 4 (the most severe response). The IRLS rating scale total score is calculated by summing the individual response scores. The highest possible score is 40, which represents the most severe RLS; the lowest possible score is 0, which represents an absence of RLS. A total of 17 participants were prematurely withdrawn from the study before Week 12.
Time Frame: Week 0 and Week 12
Population: Full Analysis Set (FAS): participants who were progressed to the treatment phase, but excluding those who did not have the target indication, those who had not received at least one dose of the investigational product, and those who did not have any measured efficacy data after initiation of the study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ropinirole IR-Ropinirole IR: Participants received immediate-release (IR) tablets of ropinirole once daily for 12 weeks in the double-blind treatment period. The dose of IP was upward titrated from 0.25 milligram (mg)/day to 0.5 mg/day at an interval of at least 1 week, followed by upward titration in increments of 0.5 mg/day at intervals of at least 1 week until sufficient efficacy was obtained (targeting "much improved" or "very much improved" in the investigator/subinvestigator-assessed Clinical Global Impression - Improvement [CGI-I]) without a safety/tolerability problem, although the dose did not exceed 3 mg/day. All participants completing the double-blind treatment period were eligible to continue in the open-label long-term treatment period. In the open-label period, participants were to receive ropinirole IR tablets once daily for 52 weeks with a similar upward titration method as in the double-blind treatment period.
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 22 | 12
units on a scale
  Week 0, n=22, 12 | 26.0 (5.51) | 24.0 (3.64)
  Week 12, n=12, 5 | 15.9 (9.97) | 9.2 (5.26)

2. Secondary Outcome: IRLS Rating Scale Total Score for Participants Who Withdrew in the Long-term Treatment Period (LONG WD)
Description: The IRLS rating scale is an investigator-rated scale consisting of 10 questions with a choice of 5 responses each. These responses are numerically scored from 0 (the least severe response) to 4 (the most severe response). The IRLS rating scale total score is calculated by summing the individual response scores. The highest possible score is 40, which represents the most severe RLS; the lowest possible score is 0, which represents an absence of RLS.
Time Frame: LONG WD (up to Week 64)
Population: FAS. One participant in each group had no measurement data and thus was not included in the analysis. These two participants were withdrawn from the study without receiving the IP in the long-term treatment period.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ropinirole IR-Ropinirole IR: Participants received ropinirole IR tablets once daily for 12 weeks in the double-blind treatment period. The dose of IP was upward titrated from 0.25 mg/day to 0.5 mg/day at an interval of at least 1 week, followed by upward titration in increments of 0.5 mg/day at intervals of at least 1 week until sufficient efficacy was obtained (targeting "much improved" or "very much improved" in the investigator/subinvestigator-assessed CGI-I) without a safety/tolerability problem, although the dose did not exceed 3 mg/day. All participants completing the double-blind treatment period were eligible to continue in the open-label long-term treatment period. In the open-label period, participants were to receive ropinirole IR tablets once daily for 52 weeks with a similar upward titration method as in the double-blind treatment period.
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 11 | 4
units on a scale | 18.0 (12.26) | 16.5 (4.12)

3. Secondary Outcome: Number of Participants With the Indicated Clinical Global Impression-Improvement (CGI-I) Scores at Week 12
Description: The CGI-I assesses the participant's improvement or worsening of RLS from baseline with the following eight grades: 0 = Not Assessed, 1 = Very Much Improved, 2 = Much Improved, 3 = Minimally Improved, 4 = No Change, 5 = Minimally Worse, 6 = Much Worse, and 7 = Very Much Worse.
Time Frame: Week 12
Population: FAS. Participants withdrawn from the study before Week 12 were not included in the analysis.
Measure: Number; unit: participants
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 12 | 5
participants
  Not Assessed | 0 | 0
  Very Much Improved | 2 | 3
  Much Improved | 3 | 1
  Minimally Improved | 4 | 1
  No Change | 2 | 0
  Minimally Worse | 1 | 0
  Much Worse | 0 | 0
  Very Much Worse | 0 | 0

4. Secondary Outcome: Number of Participants With the Indicated CGI-I Scores for Participants Who Withdrew From the Double-Blind Treatment Period (DBT WD)
Description: as for outcome 3
Time Frame: DBT WD (up to Week 12)
Population: FAS. Participants with missing DBT WD data were not included in the analysis.
Measure: Number; unit: participants
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 8 | 7
participants
  Not Assessed | 0 | 0
  Very Much Improved | 0 | 1
  Much Improved | 3 | 2
  Minimally Improved | 2 | 3
  No Change | 2 | 0
  Minimally Worse | 0 | 0
  Much Worse | 1 | 0
  Very Much Worse | 0 | 1

5. Secondary Outcome: Number of Participants With the Indicated CGI-I Scores for Participants Who Withdrew fn the Long-term Treatment Period (LONG WD)
Description: as for outcome 3
Time Frame: LONG WD (up to Week 64)
Population: FAS. Participants with no measurement data in the long-term treatment period because of their premature withdrawal without receiving the IP in that period were not included in the analysis.
Measure: Number; unit: participants
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 11 | 4
participants
  Not Assessed | 0 | 0
  Very Much Improved | 3 | 0
  Much Improved | 1 | 2
  Minimally Improved | 4 | 2
  No Change | 0 | 0
  Minimally Worse | 3 | 0
  Much Worse | 0 | 0
  Very Much Worse | 0 | 0

6. Secondary Outcome: Johns Hopkins Restless Legs Syndrome Quality of Life (RLSQOL) Questionnaire Overall Life Impact Score at Week 0 and Week 12
Description: The RLSQOL questionnaire is a participant-rated questionnaire designed to assess the impact of RLS on the lives of participants. It consists of 18 items, 10 of which contribute to a single summary score (overall life impact). The response for each item is coded from 1 to 5, with 1 representing the best quality of life and 5 representing the worst quality of life. The lowest possible overall life impact score is 0, and the highest possible overall life impact score is 100. The score of 100 represents the best possible quality of life.
Time Frame: Week 0 and Week 12
Population: FAS. Participants withdrawn from the study before Week 12 were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 22 | 12
units on a scale
  Week 0, n=22, 12 | 77.50 (15.736) | 73.13 (10.287)
  Week 12, n=12, 5 | 85.63 (14.852) | 90.50 (7.786)

7. Primary Outcome: IRLS Rating Scale Total Score for Participants Who Withdrew From the Double-Blind Treatment Period (DBT WD)
Description: The IRLS rating scale is an investigator-rated scale consisting of 10 questions with a choice of 5 responses each. These responses are numerically scored from 0 (the least severe response) to 4 (the most severe response). The IRLS rating scale total score is calculated by summing the individual response scores. The highest possible score is 40, which represents the most severe RLS; the lowest possible score is 0, which represents an absence of RLS. A total of 17 participants were prematurely withdrawn from the study before Week 12, and 2 participants had missing DBT WD data.
Time Frame: DBT WD (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 8 | 7
units on a scale | 20.3 (10.77) | 16.3 (10.42)

8. Secondary Outcome: Johns Hopkins RLSQOL Questionnaire Overall Life Impact Score for Participants Who Withdrew From the Double-Blind Treatment Period (DBT WD)
Description: as for outcome 6
Time Frame: DBT WD (up to Week 12)
Population: FAS. Participants with missing DBT WD data were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 8 | 7
units on a scale | 75.00 (12.956) | 84.64 (9.835)

9. Secondary Outcome: Johns Hopkins RLSQOL Questionnaire Overall Life Impact Score for Participants Who Withdrew in the Long-term Treatment Period (LONG WD)
Description: as for outcome 6
Time Frame: LONG WD (up to Week 64)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 11 | 4
units on a scale | 79.32 (27.502) | 87.50 (11.365)

10. Secondary Outcome: The Pittsburgh Sleep Quality Index (PSQI) Total Score at Week 0 and Week 12
Description: The PSQI consists of the following 7 domains: sleep quality, duration getting to sleep, sleep duration, sleep adequacy, sleep disturbance, use of sleeping pill, and somnolence. These domains are numerically scored from 0 to 3, with 0 representing the least severe response and 3 representing the most severe response. The PSQI total score is calculated by summing the individual domain scores. The highest possible score is 21, which represents the most disturbances in sleep quality; the lowest possible score is 0, which represents an absence of disturbances in sleep quality.
Time Frame: Week 0 and Week 12
Population: FAS. Participants withdrawn from the study before Week 12 were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 22 | 12
units on a scale
  Week 0, n=22, 12 | 10.3 (2.98) | 10.5 (3.71)
  Week 12, n=12, 5 | 7.3 (2.90) | 8.6 (2.51)

11. Secondary Outcome: The PSQI Total Score for Participants Who Withdrew From the Double-Blind Treatment Period (DBT WD)
Description: as for outcome 10
Time Frame: DBT WD (up to Week 12)
Population: FAS. Participants with missing DBT WD data were not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 8 | 7
units on a scale | 7.8 (3.54) | 7.3 (3.15)

12. Secondary Outcome: The PSQI Total Score for Participants Who Withdrew fn the Long-term Treatment Period (LONG WD)
Description: as for outcome 10
Time Frame: LONG WD (up to Week 64)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 11 | 4
units on a scale | 8.8 (3.57) | 9.3 (3.10)

13. Secondary Outcome: Number of Participants With the Indicated Responses to the Patient Satisfaction Question at Week 0 and Week 12
Description: Participants responded to a question about their satisfaction with the IP on the following 1 to 7 scale: 1 = very much satisfied; 2 = satisfied; 3 = somewhat satisfied; 4 = neither satisfied nor dissatisfied; 5 = somewhat dissatisfied; 6 = dissatisfied; and 7 = very dissatisfied. At Week 0, participants responded to a question about their satisfaction with their prior medications.
Time Frame: Week 0 and Week 12
Population: FAS. Participants withdrawn from the study before Week 12 were not included in the analysis.
Measure: Number; unit: participants
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 22 | 12
participants
  Week 0, n=22,12; Very satisfied | 0 | 1
  Week 0, n=22, 12; Satisfied | 3 | 6
  Week 0, n=22, 12; Somewhat satisfied | 4 | 2
  Week 0, n=22, 12; Neither satisfied/dissatisfied | 10 | 2
  Week 0, n=22, 12; Somewhat dissatisfied | 1 | 1
  Week 0, n=22, 12; Dissatisfied | 3 | 0
  Week 0, n=22, 12; Very dissatisfied | 1 | 0
  Week 12, n=12, 5; Very satisfied | 0 | 0
  Week 12, n=12, 5; Satisfied | 4 | 3
  Week 12, n=12, 5; Somewhat satisfied | 0 | 1
  Week 12, n=12, 5; Neither satisfied/dissatisfied | 3 | 1
  Week 12, n=12, 5; Somewhat dissatisfied | 1 | 0
  Week 12, n=12, 5; Dissatisfied | 3 | 0
  Week 12, n=12, 5, Very dissatisfied | 1 | 0

14. Secondary Outcome: Number of Participants With the Indicated Responses to the Patient Satisfaction Question for Participants Who Withdrew fn the Long-term Treatment Period (LONG WD)
Description: as for outcome 13
Time Frame: LONG WD (up to Week 64)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 11 | 4
participants
  Very satisfied | 0 | 1
  Satisfied | 2 | 0
  Somewhat satisfied | 3 | 1
  Neither satisfied/dissatisfied | 2 | 1
  Somewhat dissatisfied | 0 | 1
  Dissatisfied | 2 | 0
  Very dissatisfied | 2 | 0

15. Secondary Outcome: Number of Participants With the Indicated Responses to the Patient Satisfaction Question for Participants Who Withdrew From the Double-Blind Treatment Period (DBT WD)
Description: as for outcome 13
Time Frame: DBT WD (up to Week 12)
Population: FAS. Participants with missing DBT WD data were not included in the analysis.
Measure: Number; unit: participants
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 8 | 7
participants
  Very satisfied | 2 | 2
  Satisfied | 0 | 1
  Somewhat satisfied | 1 | 0
  Neither satisfied/dissatisfied | 3 | 2
  Somewhat dissatisfied | 1 | 1
  Dissatisfied | 0 | 0
  Very dissatisfied | 1 | 1

16. Secondary Outcome: Mean Daily Number of Hours of RLS Symptoms by Timeframe at Week 0 and Week 12
Description: Participants recorded the onset time and total duration of RLS symptoms on their diary cards for 7 days from one week before each visit. Timeframes were defined as follows: daytime, 7:00AM to 4:59PM; evening, 5:00PM to 7:59PM; and nighttime, 8:00PM to 6:59AM.
Time Frame: Week 0 and Week 12
Population: FAS. Participants without symptoms were not included in the analysis of Week 0 data. Participants without symptoms and participants prematurely withdrawn from the study were not included in the analysis of Week 12 data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 21 | 12
hours
  Daytime, Week 0, n=16, 9 | 1.794 (1.6875) | 1.857 (1.9437)
  Daytime, Week 12, n=7, 3 | 1.482 (1.3927) | 0.735 (0.3841)
  Evening, Week 0, n=11, 9 | 1.296 (0.7910) | 1.148 (0.8170)
  Evening, Week 12, n=6, 2 | 1.097 (0.9323) | 0.783 (0.3064)
  Nighttime, Week 0, n=21, 12 | 2.256 (1.5310) | 2.318 (2.3618)
  Nighttime, Week 12, n=9, 4 | 1.726 (1.4537) | 1.688 (1.1607)

17. Secondary Outcome: Mean Daily Number of Hours of RLS Symptoms by Timeframe for Participants Who Withdrew From the Double-Blind Treatment Period (DBT WD)
Description: as for outcome 16
Time Frame: DBT WD (up to Week 12)
Population: FAS. Only participants with symptoms who were able to record them in the diary card were included in the analyses of the DBT WD data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 3 | 2
hours
  Daytime, n=1, 2 | 9.590 (NA) — Only one participant was analyzed in this group at this time point. | 2.900 (3.6770)
  Evening, n=1, 1 | 2.590 (NA) — Only one participant was analyzed in this group at this time point. | 2.590 (NA) — Only one participant was analyzed in this group at this time point.
  Nighttime, n=3, 2 | 1.802 (2.7692) | 2.936 (3.1422)

18. Secondary Outcome: Mean Daily Number of Hours of RLS Symptoms by Timeframe for Participants Who Withdrew fn the Long-term Treatment Period (LONG WD)
Description: as for outcome 16
Time Frame: LONG WD (up to Week 64)
Population: FAS. Only participants with symptoms who were able to record them in the diary card were included in the analyses of the and LONG WD data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 2 | 2
hours
  Daytime, n=0, 2 | NA (NA) — No participants were analyzed in this group at this time point. | 0.883 (0.7778)
  Evening, n=1, 2 | 0.200 (NA) — Only one participant was analyzed in this group at this time point. | 1.948 (0.6399)
  Nighttime, n=2, 1 | 2.432 (2.9446) | 0.867 (NA) — Only one participant was analyzed in this group at this time point.

19. Secondary Outcome: Drug Clearance Rate On-Dialysis and Off-Dialysis During the Maintenance Dose Treatment Phase (in the Long-term Treatment Period)
Description: For on-dialysis analysis, measurements were to have been taken 1 hour before dialysis, in the artery/vein at the beginning, during, and end of dialysis, and 1 hour after dialysis. For off-dialysis analysis, measurements were to have been taken 1 hour before dialysis, at the beginning, during, and end of dialysis, and 1 hour after dialysis.
Time Frame: Week 12 through Week 64
Population: PK analysis was not performed because there were no participants (who had received a maintenance dose of the IP for more than 1 week in the long-term treatment period) from whom a blood sample could be collected when decision of study termination was made.
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were to be collected from the start of the IP (Week 0) through Week 64 and during the 4-week follow-up period. The maximum observed duration of exposure to the IP was 168 days because of the early termination of the study.
Arm/Group | Ropinirole IR-Ropinirole IR | Placebo-Ropinirole IR
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/12
Other Adverse Events (participants affected / at risk) | 16/22 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole IR-Ropinirole IR (N=22) | Placebo-Ropinirole IR (N=12)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole IR-Ropinirole IR (N=22) | Placebo-Ropinirole IR (N=12)
Nasopharyngitis (Infections and infestations) | 9 | 6
Gastroenteritis (Infections and infestations) | 2 | 0
Hordeolum (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.